CLINICAL TRIAL: NCT06057493
Title: Analytic Validation of the Optina Retinal Deep Phenotyping.TM (RDP) Platform
Brief Title: RDP Reliability Study
Status: Completed | Type: Observational
Sponsor: Optina Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-008
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retinal Imaging with Optina4C Camera — The study consists of 2 visits and 8 Imaging sessions:
  The participant will go through four (8) imaging sessions in two visits with the Optina-4CTM cameras to get pictures of your retina. These imaging sessions will be done by three qualified operators who have been trained on the study device by Optina Diagnostics.

SUMMARY:
This is an observational study designed to assess the reliability and consistency of the Optina awAIrTM CAS Test for detecting phenotypic changes in the retina that are associated with beta-amyloid status (positive or negative). The purpose of this study is to ensure that the retinal image capture process is consistent and under control, regardless of the operator or the time of measurement. The study will include enough repeated measurements on different systems, by three operators, and at different times to demonstrate.

DETAILED DESCRIPTION:
The purpose of this study is to assess the reliability of the Optina Retinal Deep Phenotyping.TM(RDP) platform. The RDP Platform is comprised of the Optina-4CTM retinal camera and its Optina-4C ConnectTM software, as well as the Optina awAIrTM-CAS Test (also called CAS Test) for detecting phenotypic changes in the retina that are associated with cerebral beta-amyloid status (positive or negative). This study will quantify points of variability in the data input for the CAS Test, including:

* Left eye vs. right eye (retinal scan)
* Eye algorithm selection (eye assessment obtained from different eye specialists either an Ophthalmologist or an Optometrist)
* Hardware variability (Inter-instrument Variability retinal scans obtained from different Optina-4CTM cameras)
* Inter-operator variability (retinal scans obtained from different Users of the Optina-4CTM camera)
* Intra-operator variability (retinal scans obtained by the same user on the same Optina-4CTM camera

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 50 years and older with vision in both eyes.
* Sufficient fluency in English or French to participate in study visits.
* Ability to give informed consent.
* Individuals with both eyes meet the eligibility criteria for retinal imaging.

Exclusion Criteria:

* Pupil dilation contraindicated (due to pathology, or presence of 3 quadrants with Van Herick grading of 0 or 1 without iridotomy).
* Inadequate pupil dilatation (< 6mm diameter) preventing uniform illumination of the retina with the Optina 4CTM camera.
* Diagnosis of glaucoma or signs of glaucoma (excavation ratio ≥0.7).
* Signs of vascular occlusion or retinopathy (microaneurysm, exudate, hemorrhage, or edema) within a diameter of 10 mm from the mid-point between the optic nerve head and the macula.
* Presence of drusen and/or age-related macular degeneration (AREDS 9-step scale

  ≥4 - cumulative drusen area diameter ≥ 250 µm, pigmentary changes and cumulative drusen area diameter ≥ 63 µm or pigmentary changes and cumulative geographic atrophy area diameter ≥ 354 µm).
* Nuclear sclerosis > 2 (LOCS II four-point grading system) or presence of central cortical or central posterior subcapsular cataract.
* Deficient visual fixation (inability to fixate for at least 2 s).
* Refractive error outside the range of -15 D to +15 D.
* Corneal or media opacities (e.g., Weiss ring) affecting retinal imaging on a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula (i.e., the area of interest for the Optina 4CTM imaging)
* Scar, atrophy, naevus, tumor, epiretinal membrane or retinal pucker with a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula.
* Papilledema and/or optic disc swelling.
* Macular anomaly (e.g., macular hole, dystrophy, degeneration).
* Inability to obtain up to 5 images or a minimum of 3 images of satisfactory quality with the Optina 4CTM per the Optina Diagnostics quality index software and /or per the eye specialists' evaluation. This exclusion criterion also applies if participants are unable to provide the required number of images during the second visit as well.
* Currently taking or has previously taken cerebral amyloid modifying medication.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women 50 years and older who can undergo pupil dilation for both eyes and are not contraindicated for mydriatic imaging with a fundus camera.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
The reliability of the investigational device's imaging process will be analyzed using agreement of CAS Test results within 95% confidence intervals for the following conditions: | 12 months
  * Eye to eye variability
  * Eye selection process variability
  * Instrument to instrument variability
  * Inter-Operator variability
  * Intra-Operator variability

CONTACTS AND LOCATIONS:
Overall Officials: Ramina Nissan, O.D, Principal Investigator — LMC Montreal Ville
Locations (1):
- LMC Montreal Ville St Laurent, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No